CLINICAL TRIAL: NCT07071233
Title: Efficacy of Vitamin C Supplementation on Serum TNF-α Levels and Disease Activity in Systemic Lupus Erythematosus Patients
Brief Title: Efficacy of Vitamin C Supplementation on Serum TNF-α Levels and Disease Activity in SLE Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Sriwijaya (Other)
Responsible Party: Principal Investigator, Yuniza, Principal investigator, Division of Allergy Immunology Faculty Member, Department of Internal Medicine, Universitas Sriwijaya/Mohammad Hoesin General Hospital, Universitas Sriwijaya
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 04.03DXVIII0608ETIK204/2024
Record Dates: First submitted 2025-06-30; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Systemic Lupus Erythematosus (SLE)
Keywords: systemic lupus erythematosus; SLE; vitamin c; TNF-alpha; Mex-SLEDAI; disease activity
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: The study was The study was designed as a single-center double-blind randomized controlled clinical trial. Participants were randomized into two groups receiving Vitamin C or placebo
Who Masked: Participant, Care Provider, Investigator
Masking Description: Triple (Participant, Care Provider, Investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin C (Experimental): The patients were given a tablet containing Vitamin C 500 mg twice a day
  Interventions: Dietary Supplement: Vitamin C
- Placebo (Placebo Comparator): The patients were given a placebo capsule with a similar color, shape, size and taste twice a day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin C — The patients received vitamin C supplementation
  Arms: Vitamin C
Dietary Supplement: Placebo — Patients received placebo capsules
  Arms: Placebo

SUMMARY:
The study aimed to evaluate the efficacy of vitamin C supplementation compared to placebo towards TNF-α levels and disease activity with the MEX-SLEDAI score in Systemic Lupus Erythematosus (SLE) patients. The current study was designed as a single-center double-blind randomized controlled clinical trial. The participants were voluntarily recruited ≥ 18 years old SLE patients, with mild to moderate disease activity and did not consumed vitamin C 1 week prior to the trial study. Participants were randomized into two groups receiving vitamin C supplementation, or placebo. TNF-α levels and MEX-SLEDAI score were evaluated at the beginning and at the end of the 8 week trial for analysis.

ELIGIBILITY:
Inclusion Criteria:

1. All patients diagnosed with systemic lupus erythematosus with mild-moderate disease activity who are treated at the Allergy-Immunology Department of RSMH.
2. Patients aged over 18 years.
3. Willing to participate in the study by signing an informed consent form.

Exclusion Criteria

1. Pregnant or breastfeeding.
2. Patients with other immune disorders such as HIV, Rheumatoid Arthritis, Pulmonary Tuberculosis, chronic liver disease, and malignancies.
3. Patients currently taking supplements containing vitamin C for more than 1 week.
4. Patients with a diagnosis of SLE with severe disease activity or those who have reached remission.
5. Patients who are hospitalized due to SLE.
6. Patients with comorbid conditions such as hemochromatosis and gastritis.

Drop-out Criteria

1. Patients who discontinue vitamin C for more than 3 weeks.
2. Death.
3. Development of serious drug side effects, requiring discontinuation of the medication.
4. Patients who are readmitted or experience symptom deterioration during the intervention period.
5. Loss to follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
MEX-SLEDAI score | From enrollment to the end of the treatment at 8 weeks
  To determine the effectiveness of adding vitamin C compared to placebo towards disease activity in SLE patients, measured with MEX-SLEDAI score
TNF-α | From enrollment to the end of the treatment at 8 weeks
  To determine the effectiveness of adding vitamin C compared to placebo towards TNF-α levels concentration change in SLE patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Mohammad Hoesin General Hospital, Palembang, South Sumatera, Indonesia

REFERENCES:
- [Background] Kong EH, Ma SY, Jeong JY, Kim KH. Effects of L-ascorbic acid on the production of pro-inflammatory and anti-inflammatory cytokines in C57BL/6 mouse splenocytes. KMJ. 2015 Jan 20;30(1):41-9.
- [Background] Islam MA, Khandker SS, Kotyla PJ, Hassan R. Immunomodulatory Effects of Diet and Nutrients in Systemic Lupus Erythematosus (SLE): A Systematic Review. Front Immunol. 2020 Jul 22;11:1477. doi: 10.3389/fimmu.2020.01477. eCollection 2020. PMID 32793202